CLINICAL TRIAL: NCT00190957
Title: Atomoxetine Treatment of Adults With ADHD and Comorbid Alcohol Abuse: A Randomized, Placebo-Controlled Trial
Brief Title: Atomoxetine Treatment of Adults With ADHD and Comorbid Alcohol Abuse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7069; B4Z-MC-LYBY
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: ADHD; Comorbid Alcohol Abuse
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine
Drug: placebo

SUMMARY:
Atomoxetine Treatment of Adults with ADHD and Comorbid Alcohol Abuse

ELIGIBILITY:
Inclusion Criteria:

You must be at least 18 years old.

You must have a diagnosis of ADHD and a diagnosis of alcohol abuse or dependence.

You must have acceptable results on blood and urine tests and an electrocardiogram (ECG).

Your recent drinking history must meet specific requirements.

Exclusion Criteria:

You have taken atomoxetine in the past.

You have a psychiatric disorder, other than ADHD and alcohol abuse or dependence, for which you will need psychiatric medication.

You have cognitive impairment (such as memory loss), a brain injury, or a seizure disorder.

You have a history of severe allergies to more than 1 class of medication or multiple bad reaction to drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2004-08; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To test that atomoxetine is superior to placebo in reducing ADHD severity as measured by the Adult ADHD Investigator Symptom Rating Scale (AISRS) Total score and is superior to placebo in time to relapse of alcohol abuse at 12 weeks.

SECONDARY OUTCOMES:
Total alcohol consumption (mean drinks/day) during the final week of treatment is lower in patients treated with atomoxetine than in patients receiving placebo.
The proportion of drinking days is smaller for atomoxetine-treated patients compared with those in the placebo group.
Time to relapse of alcohol abuse is longer for atomoxetine-treated patients compared with those in the placebo group.
Number of drinks per drinking day is smaller for patients treated with atomoxetine compared with placebo.
The proportion of substance use days, for substances other than alcohol, is smaller among patients treated with atomoxetine as compared with placebo.
After approximately 12 weeks of treatment, patients who receive atomoxetine will have superior social and occupational functioning compared with those who receive placebo as assessed by changes in the EWPS.
Global functioning as assessed by the CGI-Overall-S and the CGI-I are superior in patients treated with atomoxetine as compared with those treated with placebo.
Improvement in depressive symptoms as assessed by the HAM-D-17.
Improvement in anxiety symptoms as assessed by the HAM-A.
Improvement in self-reported ADHD symptoms as assessed by the ASRS.
Improvement in self-rated symptoms of alcohol cravings as assessed by the OCDS.
Improvement in specific symptoms of ADHD as assessed by the WRAADDS.
Improvement in the self-rated adaptive functioning as assessed by the ASR.
Improvement in the informant-related adaptive functioning as assessed by the ABCL.
Improvement in work, social, and home life functioning as assessed by the Sheehan Disability Scale.
Improvement in general quality of life as assessed by the SF-36 Health Status Survey and the Q-LES-Q-SF.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, El Centro, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Poway, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New London, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cambridge, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Okemos, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moorestown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Middleton, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Vancouver, Canada

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] Wilens TE, Adler LA, Tanaka Y, Xiao F, D'Souza DN, Gutkin SW, Upadhyaya HP. Correlates of alcohol use in adults with ADHD and comorbid alcohol use disorders: exploratory analysis of a placebo-controlled trial of atomoxetine. Curr Med Res Opin. 2011 Dec;27(12):2309-20. doi: 10.1185/03007995.2011.628648. Epub 2011 Oct 27. PMID 22029549
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com